CLINICAL TRIAL: NCT06344962
Title: Comparison of Clinical Effects of Absorbable and Non-absorbable Suture in Bronchial Sleeve Resection
Brief Title: Clinical Effects of Absorbable and Non-absorbable Suture in Bronchial Sleeve Resection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, jiaowenjie, Professor, The Affiliated Hospital of Qingdao University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QYFYKYLL930611921
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Suture, Complication
Keywords: Suture; Bronchial Sleeve Resection; Central Primary Lung Cancer; Non-Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Absorbable Suture Group (Experimental): All enrolled patients will accept bronchial sleeve resection and lymphadenectomy. If fast-frozen pathology of the resection margin of bronchus confirms negative, We will use the absorbable sutures for bronchial anastomosis.
  Interventions: Device: Absorbable Suture
- Non-absorbable Suture Group (Experimental): All enrolled patients will accept bronchial sleeve resection and lymphadenectomy. If fast-frozen pathology of the resection margin of bronchus confirms negative, We will use the non-absorbable sutures for bronchial anastomosis.
  Interventions: Device: Non-absorbable Suture

INTERVENTIONS:
Device: Absorbable Suture — 3-0 V-Loc
  Arms: Absorbable Suture Group
Device: Non-absorbable Suture — 3-0 Prolene
  Arms: Non-absorbable Suture Group

SUMMARY:
Bronchial sleeve resection is performed as an alternative to pneumonectomy for lung cancer patients with centrally located lesions and limited cardiopulmonary reserve. Intraoperative bronchial anastomosis is very complex and difficult, mainly due to the difficulty of suturing and knotting in limited space. There are currently few studies comparing the clinical effects of absorbable and non-absorbable suture in bronchial sleeve resection. So the investigator wants to conduct a prospective study, trying to figure out this problem.

DETAILED DESCRIPTION:
Lung cancer has been one of the most serious life-threatening diseases of human society. It has the highest morbidity and mortality worldwide among all the malignant tumors. Although the treatment of lung cancer is increasingly diverse, surgical resection is still the mainstay.

Pneumonectomy, as a surgical approach for central primary lung cancer, is very harmful to patients. Bronchial sleeve resection is performed as an alternative to pneumonectomy for lung cancer patients with centrally located lesions and limited cardiopulmonary reserve. Intraoperative bronchial anastomosis is very complex and difficult, mainly due to the difficulty of suturing and knotting in limited space. Both absorbable and non-absorbable suture are used for it. But there are currently few studies comparing the clinical effects of absorbable and non-absorbable suture in bronchial sleeve resection. So the investigator wants to conduct a prospective study, trying to figure out this problem.

The investigator sets incidence rate of anastomotic complications as the primary endpoint. According to the calculation, a total of 40 patients will be enrolled (each group has 20 patients).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years old.
2. The tumor is located in the opening of bronchus, or the edge of the tumor is less than 2 cm away from the opening of the bronchi, while the distance between the edge of the tumor and the carina is more than 1.5 cm.
3. Patients with pathological diagnosis of non-small cell lung cancer.
4. No distant metastasis in preoperative clinical evaluation.
5. Adequate cardiac function, pulmonary function, liver function and renal function for anesthesia and bronchial sleeve resection.
6. American Society of Anesthesiologists (ASA) score: Grade I-III.
7. Patients who can coordinate the treatment and research and sign the informed consent.

Exclusion Criteria:

1. Patients with a significant medical condition which is thought unlikely to tolerate the surgery or unsuitable for this study after the evaluation of the investigator.
2. Patients with psychiatric disease who are expected lack of compliance with the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of anastomotic complications | 12 months after surgery
  such as anastomotic stenosis, anastomotic fistula and so on

SECONDARY OUTCOMES:
Time of bronchial anastomosis | During surgery
  From the first stitch to the last stitch
Number of stitches | During surgery
  During bronchial anastomosis
5-year survival rate | 5 years after surgery
  Follow up for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Wenjie Jiao, PhD, Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- the Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No